CLINICAL TRIAL: NCT06934915
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Groups Trial of Prednisone in Adults With an Immune-Mediated Subtype of Autism Spectrum Disorder
Brief Title: Prednisone in Adults With an Immune-Mediated Subtype of Autism Spectrum Disorder
Acronym: PREDICT
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Christopher John McDougle, M.D. (Other)
Responsible Party: Sponsor-Investigator, Christopher John McDougle, M.D., Director, Lurie Center for Autism, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024P003682
Record Dates: First submitted 2025-04-03; First posted 2025-04-18 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder; Autism Spectrum Disorders; Autism
Keywords: Autism Spectrum Disorder; Autistic Disorder; Autism; Autoimmunity; Autoimmune Disorders; Inflammation; Neuroinflammation; Anti-Inflammatory Agents; Corticosteroids; Glucocorticoids; Prednisone
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Autoimmune Diseases; Inflammation; Neuroinflammatory Diseases | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to prednisone or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, parents/legal guardians (i.e., study partners), site staff (including investigators), and outcomes assessors will be masked for the duration of the study. Investigative pharmacists (or designees) will be unmasked for randomization and treatment allocation. Emergency unmasking may occur at any time throughout the study in the event that knowledge of the actual treatment is absolutely essential for further management of the participant, to fulfill expedited reporting requirements, or if requested by the Data Safety and Monitoring Board (DSMB).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisone (Experimental): Eligible participants will receive prednisone for up to 16 weeks. The treatment period consists of 3 structured phases: Dose Escalation (Weeks 1-5), Optimal Dose Maintenance (Weeks 6-10), and Gradual Dose Reduction (Weeks 11-16).
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): Eligible participants will receive a matching placebo for up to 16 weeks. The treatment period consists of 3 structured phases: Dose Escalation (Weeks 1-5), Optimal Dose Maintenance (Weeks 6-10), and Gradual Dose Reduction (Weeks 11-16).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — Starting dose: 5 mg daily. Maximum dose: 60 mg daily. Dosage forms: 5 mg, 10 mg, and 20 mg capsules.
  Arms: Prednisone
Drug: Placebo — Capsules identical in size and appearance to those containing prednisone. Placebo capsules contain inactive ingredients.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn how prednisone affects adults with autism spectrum disorder (ASD). It will also learn about the safety of prednisone. The main questions it aims to answer are:

* How does prednisone affect the core features and associated target symptoms of ASD in adults with an immune-mediated subtype of ASD?
* Is prednisone safe for autistic adults without causing too many side effects?
* Does this study warrant larger trials studying anti-inflammatory drugs in this subject population?

Researchers will compare the drug prednisone to a placebo (a look-alike substance that contains no drug) to see how prednisone affects autistic adult males.

Participants will:

* Visit the clinic 2 times for a screening and baseline visit.
* Take prednisone or a placebo every day for 16 weeks.
* Visit the clinic 2 times for checkups, tests, questionnaires, and dose changes, and 1 time for a follow-up visit 4 weeks after stopping the study drug.
* Provide blood and urine samples for testing up to 4 times.
* Complete 8 remote calls every 1-2 weeks for checkups and dose changes.
* Keep a diary of the dose and times they take the study drug every day and any symptoms or side effects they experience.

DETAILED DESCRIPTION:
* Randomized, double-blind, placebo-controlled, parallel-groups, flexibly dosed trial. Eligible autistic male participants will be randomized 1:1 to receive prednisone or a placebo.
* Participants will attend up to 5 in-person study visits: screening, baseline, Week 5, Week 10, and Week 20 (post-discontinuation follow-up).
* Interim dose adjustments will be determined during 8 scheduled remote visits: Weeks 1-4, Week 7, Week 12, Week 14, and Week 16.
* Blood and urine specimens will be collected for safety and biomarker assessments: screening, Week 5, Week 10, and Week 20.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 50 years of age (inclusive) and assigned male at birth.
2. Diagnostic Statistical Manual of Mental Disorders (DSM), Fourth Edition, Text Revision (DSM-IV-TR) diagnosed autistic disorder, and DSM, Fifth Edition, Text Revision (DSM-5-TR) diagnosed autism spectrum disorder (ASD), level 2 or 3. A qualified (board-eligible or board-certified) psychiatrist or psychologist, with experience in diagnostic determinations of ASD, will make a final diagnostic determination based on clinical history, clinical observations, medical records, mental status exams, and screening measures.
3. A Clinical Global Impression-Severity (CGI-S) rating ≥ 4 ("Moderate") at screening (and baseline).
4. A non-verbal IQ in the range of moderate intellectual disability or higher (≥ 35), as measured by the non-verbal Abbreviated IQ (ABIQ) score of the Stanford-Binet Intelligence Scales, Fifth Edition (SB-5), or mental age of at least 18 months, as measured by the Cognitive and Adaptive Behavior subscales of the Developmental Profile (DP-4) Parent/Caregiver Interview form.
5. Participation of a study partner who has consistent contact with the participant and is willing and able to attend visits, oversee the participant's compliance with the protocol and study medication, and report on the participant's status through study assessments.
6. Participant reports ≥ 1 of the following:

   * A diagnosed comorbid autoimmune disease (e.g., Crohn's disease, Graves' disease, Hashimoto's disease, psoriasis, rheumatoid arthritis, ulcerative colitis, type 1 diabetes mellitus, etc.).
   * Current biomarker evidence of critical indicators of inflammation/autoimmunity, such as elevated levels of C-reactive protein (CRP) or abnormal value of antinuclear antibodies (ANA).
   * A significant family history of autoimmunity, defined as having ≥ 1 first-degree relative or ≥ 2 second-degree relatives with autoimmune diseases. The Principal Investigator (PI) will make the final determination on this criterion.
7. Participant reports a history of ≥ 2 of the following conditions or complaints:

   * Gastrointestinal symptoms
   * Epilepsy or seizures
   * Ear tube placements
   * Sleep disorder or difficulty sleeping
8. Any concomitant medications or interventions for ASD-related symptoms (e.g., alpha-2 agonists, anticonvulsants, antidepressants, antipsychotics, anxiolytics, gastrointestinal medications, medications for sleep disorders, probiotics, stimulants, behavioral therapies, psychosocial interventions, speech therapy, etc.) have been stable for at least 4 weeks prior to the screening visit and the participant/study partner intend to maintain a stable regimen throughout the trial.
9. Participant can tolerate swallowing large capsules.
10. Participant is willing and able, in the investigator's opinion, to comply with all study procedures.

Individuals must satisfy the following criteria to be enrolled as study partners:

1. The study partner is fluent in English.
2. The study partner is a caregiver or an individual who has consistent contact with the participant, knows the participant well, and is willing and able to attend visits, oversee the participant's compliance with the protocol and study medication, and report on the participant's status through study assessments. The PI will make the final determination on this criterion.

Exclusion Criteria:

1. DSM-5-TR diagnosed ASD, level 1, or presence of another DSM-IV-TR diagnosed pervasive developmental disorder, such as Asperger's disorder, childhood disintegrative disorder, Rett syndrome, or pervasive developmental disorder not otherwise specified (PDD-NOS). A qualified psychiatrist or psychologist will make a diagnostic determination after reviewing clinical history, clinical observations, medical records, mental status exams, and screening measures.
2. A CGI-S rating < 4 at screening (or baseline).
3. A non-verbal IQ in the range of severe or profound intellectual disability (< 35), as measured by the non-verbal ABIQ score of the SB-5, or mental age below 18 months, as measured by the Cognitive and Adaptive Behavior subscales of the DP-4 Parent/Caregiver Interview form. Individuals testing below 18 months may be enrolled after a case review by the PI and study psychologist, especially if testing scores were likely underestimated due to uncooperative behavior.
4. Previous documentation of a prolonged electroencephalogram (EEG) suggestive of Landau-Kleffner syndrome or continuous spike and wave during sleep (CSWS) syndrome.
5. Presence of a defined genetic disorder, such as Angelman syndrome, Fragile X syndrome, Noonan syndrome, Tuberous sclerosis, Williams syndrome, or any documented chromosomal or genetic abnormality with proven clinical significance in the etiology of ASD.
6. Documented significant pre- or post-natal central nervous system insult, such as an in-utero cerebral vascular accident, that is believed to have significantly contributed to the development of the individual's ASD.
7. Mitochondrial disorder verified by skin and/or muscle biopsy.
8. History of bipolar disorder or psychotic disorder, including major depressive disorder with psychotic features, schizoaffective disorder, or schizophrenia. History of a significant and interfering comorbid major psychiatric disorder, including obsessive-compulsive disorder, post-traumatic stress disorder, or substance use disorder requiring > 1 psychiatric hospitalization for treatment of specific comorbid psychiatric disorders above and beyond target symptoms associated with ASD, such as aggression, irritability, self-injury, property destruction, mood swings, or severe tantrums. Minor psychiatric disorders, such as adjustment disorder, attention-deficit hyperactivity disorder, generalized anxiety disorder, major depressive disorder, persistent depressive disorder, or social anxiety disorder, may not exclude participation. The PI will make the final determination on this exclusion criterion.
9. Concomitant medications or interventions for ASD-related symptoms (e.g., alpha-2 agonists, anticonvulsants, antidepressants, antipsychotics, anxiolytics, gastrointestinal medications, medications for sleep disorders, probiotics, stimulants, behavioral therapies, psychosocial interventions, speech therapy, etc.) have not been stable for at least 4 weeks prior to the screening visit.
10. An active bacterial, fungal, helminthic, protozoan, or viral infection that could be exacerbated by a course of prednisone, as determined by the PI.
11. Significant medical findings from history, physical examination, or laboratory testing that may be incompatible with prednisone use (e.g., participants with chronic infectious conditions or unstable diabetes mellitus).
12. Individuals with a history of seizures being treated with an anticonvulsant may be eligible if seizure-free for at least 6 months and the anticonvulsant dose has been stable for at least 4 weeks prior to the screening visit.
13. Use of immunosuppressive agents within the 6 months prior to the screening visit or concurrent use of immunosuppressive agents that, in the judgment of the PI, would interfere with study outcomes or pose unreasonable risk with prednisone administration.
14. A known hypersensitivity to prednisone or any other component of the study product.
15. The participant is deemed unsuitable for any reason by the PI, including an inability to complete or comply with study requirements.

Individuals may be excluded from enrollment as study partners if either of the following criteria are met:

1. The study partner is not fluent in English.
2. The study partner is deemed unsuitable for any reason by the PI, including an inability to complete or comply with study requirements.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-11 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Mean difference in Clinical Global Impressions-Improvement (CGI-I) ratings between the prednisone and placebo groups at Visit 9 | Baseline to Week 10
  Mean difference in CGI-I ratings between the prednisone and placebo groups at Visit 9 (efficacy). The CGI-I is a single-item measure of global symptomatic improvement compared to baseline. Improvement is rated on a 7-point scale, ranging from 1 ("Very much improved") to 7 ("Very much worse"). A global domain score of 1 ("Very much improved") or 2 ("Much improved") on the CGI-I scale will constitute a positive treatment response.

SECONDARY OUTCOMES:
Number of randomized study participants | At Baseline
  Number of randomized study participants (feasibility).
Percent of participants enrolled at Visit 9 (Week 10) and contributing a visit 9 CGI-I rating | Baseline to Week 10
  Percent of participants enrolled at Visit 9 (Week 10) and contributing a visit 9 CGI-I rating, irrespective of treatment continuation (feasibility).
Percent of participants randomized to prednisone experiencing serious adverse events (SAEs) probably or definitely related to medication | Baseline to Week 20
  Percent of participants randomized to prednisone experiencing serious adverse events (SAEs) probably or definitely related to medication (safety).
Percent of participants randomized to prednisone who complete a ten-week course of study drug | Baseline to Week 10
  Percent of participants randomized to prednisone who complete a ten-week course of study drug (tolerability).

OTHER OUTCOMES:
Change in Aberrant Behavior Checklist-Community (ABC-C) Score | Baseline to Week 10
  Change in Aberrant Behavior Checklist-Community (ABC-C) scores from Baseline to Week 10. The ABC-C is a 58-item, informant-based scale measuring psychiatric symptoms and behavioral disturbance across five domains (subscales) within the past 28 days: hyperactivity, inappropriate speech, irritability, social withdrawal/lethargy, and stereotypic behaviors. Each item is rated from 0 ("Not a problem") to 3 ("Severe problem").

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J McDougle, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Lurie Center for Autism, Lexington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to externally share IPD at this time, due to concerns regarding participant privacy, the risk of reidentification given the small and vulnerable study population, and limitations in the consent materials and protocol, which do not currently permit external data sharing. Institutional policy requires specific Data Use Agreements for any data sharing activity, and the study is protected by a Certificate of Confidentiality, further restricting disclosure of identifiable information. The research team may consider sharing de-identified data in the future, contingent upon publication of results and implementation of robust governance and approval mechanisms.